CLINICAL TRIAL: NCT03923465
Title: Clinical Outcomes of the Entire Papilla Preservation Technique With and Without Biomaterials in the Treatment of Isolated Intrabony Defects: A Randomised-controlled Clinical Trial
Brief Title: Entire Papilla Preservation Technique With and Without Biomaterials in the Treatment of Isolated Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Aslan Private Perio Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AslanPPC_RCT_01
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EPP with EMD+BS (Active Comparator): Using minimally invasive surgery, entire papilla preservation technique with the adjunctive use of amelogenins and bone substitutes
  Interventions: Procedure: Procedure: Periodontal surgery with entire papilla preservation (EPP) technique; Device: EMD application; Device: Bone substitutes application
- EPP without EMD+BS (Other): Using minimally invasive surgery, entire papilla preservation technique without the adjunctive use of amelogenins and bone substitutes
  Interventions: Procedure: Procedure: Periodontal surgery with entire papilla preservation (EPP) technique

INTERVENTIONS:
Procedure: Procedure: Periodontal surgery with entire papilla preservation (EPP) technique — After local anesthesia injection an modified flap is designed according to minimally invasive microsurgical techniques. After flap elevation, careful removal of granulation tissues from the periodontal defects is performed. Scaling and root planing of the involved dental roots is ensured and finally suture is placed.
Device: EMD application — Application of Pref-Gel for 2 minutes and then the application of Enamel Matrix Derivatives (EMD) on the surgically exposed root surface.
  Other Names: Amelogenins application
  Arms: EPP with EMD+BS
Device: Bone substitutes application — Following the application of EMD, filling the bone defect with bone substitutes.
  Arms: EPP with EMD+BS

SUMMARY:
The aim of this study is to investigate the clinical efficacy of entire papilla preservation technique with and without the adjunct of amelogenins (EMD) and bone substitutes.

DETAILED DESCRIPTION:
The present study is designed as a single-centre, parallel group, randomized, controlled clinical trial comparing the efficacy of EPP with or without biomaterials. Each patient will contribute with a single intrabony defect. Three months after completion of initial periodontal therapy, all the experimental sites will be accessed with the "EPP" technique (Aslan et al., 2017a) and carefully debrided. EDTA gel will be applied on the instrumented root surfaces. A combination of EMD and deproteinized bovine-derived bone substitute will be applied in the test group (EPP EMD + BS), while the control group (EPP) will not receive any regenerative biomaterial. Patients will be enrolled in a stringent maintenance programme with recalls on a weekly basis for the first month and then monthly controls for professional tooth cleaning up to 1 year. Clinical parameters will be recorded immediately before regenerative surgery (baseline) and 12 months after the regenerative periodontal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Clinical diagnosis of advanced periodontitis
* Having one isolated intrabony defect with probing depth (PD) ≥7 mm, clinical attachment level (CAL) ≥8 mm and at least 4 mm intrabony component involving predominantly the interproximal area of the affected tooth.
* Full-mouth plaque score (FMPS) ≤20%.
* Full-mouth bleeding score (FMBS) ≤20%.

Exclusion Criteria:

* Smokers
* Patients with known systemic diseases such as diabetes and cardiovascular diseases or using medications that affect periodontal tissues, pregnant or lactating women
* One-wall intrabony defects
* Defects that involve buccal and lingual sites
* Presence of inadequate endodontic treatment and/or restoration in the relevant teeth.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04-04 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) gain | 1-year
  CAL is measured as the distance between cemento-enamel junction and the tip of the periodontal probe

SECONDARY OUTCOMES:
Post-surgical discomfort | 1-week after surgery
  Post-surgical discomfort will be measured on a visual analog scale (VAS) and reported in millimeters. The subjects will be instructed to mark their level of pain on a line. The average change in discomfort level will be determined and compared between the two arms.
  A visual analogue scale (VAS) of 100 mm long will be used to evaluate the degree of discomfort (0=no pain/hardship; 100=unbearable pain/hardship).

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Aslan, DDS, PhD, Principal Investigator — Private Office Dr. Aslan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslan S, Buduneli N, Cortellini P. Entire Papilla Preservation Technique: A Novel Surgical Approach for Regenerative Treatment of Deep and Wide Intrabony Defects. Int J Periodontics Restorative Dent. 2017 Mar/Apr;37(2):227-233. doi: 10.11607/prd.2584. PMID 28196163
- [Background] Aslan S, Buduneli N, Cortellini P. Entire papilla preservation technique in the regenerative treatment of deep intrabony defects: 1-Year results. J Clin Periodontol. 2017 Sep;44(9):926-932. doi: 10.1111/jcpe.12780. Epub 2017 Aug 23. PMID 28727170
- [Derived] Aslan S, Buduneli N, Cortellini P. Clinical outcomes of the entire papilla preservation technique with and without biomaterials in the treatment of isolated intrabony defects: A randomized controlled clinical trial. J Clin Periodontol. 2020 Apr;47(4):470-478. doi: 10.1111/jcpe.13255. Epub 2020 Feb 3. PMID 31925811